CLINICAL TRIAL: NCT00035035
Title: A Phase 3 Trial of ALIMTA (LY231514, Pemetrexed) Plus GEMZAR Versus GEMZAR in Patients With Unresectable or Metastatic Cancer of the Pancreas.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5148; H3E-MC-JMES; NCT00049426 (obsolete NCT alias)
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2006-07-19 (Estimated); Status verified 2006-07

CONDITIONS: Pancreatic Neoplasms; Metastases, Neoplasm
Keywords: Pancreas; Cancer; Unresectable or Metastatic Cancer of the Pancreas; Alimta
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — Gemcitabine; Pemetrexed

INTERVENTIONS:
Drug: GEMZAR
Drug: ALIMTA

SUMMARY:
Definition: This study will compare the drug GEMZAR to a combination of GEMZAR plus ALIMTA for the treatment of cancer of the pancreas. Patients may be able to participate in this study if they have cancer in their pancreas that cannot be removed by surgery OR that has spread to a new site in their body.

ELIGIBILITY:
Inclusion Criteria:

* Pancreas cancer that cannot be removed by surgery OR that has spread to a new site in your body.
* You must have one tumor that can be physically measured or scanned by the doctor.
* You have not had any chemotherapy, immunotherapy, biologic therapy, or hormonal therapy for pancreas cancer, including 5-FU.
* You cannot have any radiation for 4 weeks before starting this study, and you cannot have radiation to the whole pelvis.

Exclusion Criteria:

* Treatment with any medication or device that has not been approved by regulatory agencies, like the FDA, at the time you enter the study.
* Documentation that the cancer has spread to your brain.
* Pregnant or breastfeeding.
* A second primary cancer.
* Unable to stop aspirin or non-steroidal anti-inflammatory agents (like ibuprofen) for 5-8 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (114):
- United States (40):
  - Huntsville, Alabama
  - Fountain Valley, California
  - Fullerton, California
  - Lancaster, California
  - Los Angeles, California
  - Pomona, California
  - Santa Rosa, California
  - Torrance, California
  - Fort Collins, Colorado
  - Hartford, Connecticut
  - Lake Worth, Florida
  - Miami, Florida
  - Chicago, Illinois
  - Decatur, Illinois
  - Harvey, Illinois
  - Indianapolis, Indiana
  - Wichita, Kansas
  - Crestview Hills, Kentucky
  - Louisville, Kentucky
  - Lafayette, Louisiana
  - Shreveport, Louisiana
  - Scarborough, Maine
  - Burlington, Massachusetts
  - Omaha, Nebraska
  - Albuquerque, New Mexico
  - New York, New York
  - Canton, Ohio
  - Cleveland, Ohio
  - Drexel Hill, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Johnson City, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - San Antonio, Texas
  - Tyler, Texas
  - Tacoma, Washington
  - Marshfield, Wisconsin
  - Milwaukee, Wisconsin
- Argentina (4):
  - Capitol Federal, Buenos Aires
  - Mendoza, Mendoza Province
  - Santa Fe, Rosario
  - Ciudad de Buenos Aires
- Australia (6):
  - Bankstown, New South Wales
  - Kingswood Penrith, New South Wales
  - Wollongong, New South Wales
  - Southport, Queensland
  - Fitzroy, Victoria
  - Frankston, Victoria
- Austria (3):
  - Innsbruck
  - Saint Veit Glan
  - Vienna
- Belgium (3):
  - Brussels
  - Ghent
  - Leuven
- Cali, Colombia
- France (7):
  - Strasbourg, Cedex
  - Lille
  - Marseille
  - Paris
  - Rennes
  - Rouen
  - Toulouse
- Germany (11):
  - Bielefeld, Nordhein-Westfalen
  - Berlin
  - Bremerhaven
  - Frankfurt
  - Kaiserslautern
  - Karlsruhe
  - Magdeburg
  - Mannheim
  - München
  - Neustadt/Suedharz
  - Stuttgart
- Greece (2):
  - Marousi, Athens
  - Ioannina
- Italy (3):
  - Genova
  - Ravenna
  - Roma
- Netherlands (5):
  - Breda
  - Enschede
  - Roermond
  - Sittard
  - The Hague
- Peru (2):
  - Chiclayo
  - Lima
- Portugal (4):
  - Lisbon
  - Porto
  - Santa Maria da Feira
  - Santarém
- Spain (5):
  - Elche, Alicante
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Santa Cruz de Tenerife, Santa Cruz De Tenerife
  - Zaragoza, Zaragoza
- Sweden (5):
  - Linköping
  - Lund
  - Malmo
  - Stockholm
  - Umeå
- Taiwan (4):
  - Taoyuan District, Kuei-Shan
  - Yungkang City, Tainan
  - Tainan
  - Taipei
- United Kingdom (6):
  - Bristol, Avon
  - Hull, East Yorkshire
  - Acton, London
  - Northwood, Middlesex
  - Belfast, Northern Ireland
  - Manchester
- Venezuela (3):
  - Valencia, Edo. Aragua
  - Estado Aragua, Maracay
  - Caracas